CLINICAL TRIAL: NCT06643871
Title: Adapted Physical Activity Program in a Enriched Environment and Virtual Reality - Connected Bike - for Patients Undergoing Antipsychotic Treatment in the Context of a First Episode of Psychosis
Brief Title: Adapted Physical Activity Program for Patients Undergoing Antipsychotic Treatment of a First Episode of Psychosis
Acronym: DYNAMO-PSY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: D23-P009
Record Dates: First submitted 2024-02-16; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-02

CONDITIONS: Schizophrenia; Psychosis; Schizo Affective Disorder; First Episode Psychosis (FEP)
Keywords: Schizophrenia; Adapted physical activity; Early Intervention; First Episode psychosis; Metabolic Syndrom
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DYNAMO-PSY program (Experimental): This is a feasibility study. Therfore, there is only one arm, the experimental one, where participants will be enrolled in the DYNAMO-PSY program.
  Interventions: Other: Adapted physical activity program involving connected bikes

INTERVENTIONS:
Other: Adapted physical activity program involving connected bikes — The treatment being studied involves a program (DYNAMO-PSY) of adapted physical activity with an enriched environment (connected bike, visualized and experienced routes in virtual reality) and is supervised, comprising (on average) two sessions per week, a total of 20 sessions to be completed over a maximum of 15 weeks. Each session will last 60 minutes and will be supervised by a case manager. They will be composed of a warm up, session on the bike (around 30 minutes of bicycling) and stretching. They will take place in an adequate room in the clinical research department of Saint Anne Hospital. The usual hygienic-dietetic care is not modified by the study and consists of the care proposed to patients of the GHU Paris Psychiatry and Neuroscience who have had a first psychotic episode and are treated primarily with medication: clinical and biological monitoring, dietary consultations, therapeutic education group concerning diet and lifestyle.

SUMMARY:
The purpose of this PILOT feasibility study is to verify the acceptability, feasibility, and compliance to the DYNAMO-PSY program among young adults treated with antipsychotics for a first episode of psychosis (FEP).

Our hypothesis is that the use of an immersive program of APA, including an EE with VR (connected bikes), will allow good observance to regular physical activity in patients treated with antipsychotics for a FEP. This regular practice of physical activity will prevent the onset of weight gain and metabolic syndrome. In addition, a positive effect on self-esteem, overall and particularly cognitive functioning, quality of life, and adherence to antipsychotic treatment can be expected.&amp;amp;amp;amp;amp;amp;#34;

DETAILED DESCRIPTION:
Introduction :

Patients suffering from schizophrenia (SCZ) (1% of the general French population) have an increased risk of cardio-metabolic morbidity and mortality, and their life expectancy is reduced by 15 years. In France, the incidence of psychotic disorders is estimated at 15,000 new cases per year among young people aged 15 to 25 years. Psychotic disorders have a significant socio-economic impact, and the emergence of these disorders represents a real break at the individual, social, and family levels. The first clinical signs of the FEP appear in adolescence or early adulthood, particularly because the brain is more vulnerable during this period to environmental risk factors such as substance use and stress.

Early intervention propose appropriate care from the first symptoms, including the introduction of antipsychotic treatment. However, we know that these treatments can lead to weight gain and metabolic syndrome, a risk factor for cardiovascular disease that can generate treatment discontinuation. Moreover, we know that neurocognitive disorders are predisposing factors not only for the development of early psychosis but also for the chronicity of a psychotic pathology.

Alternative approaches have been developed over the past decades to manage daily difficulties of patients with a FEP (e.g., cognitive issues, symptoms, metabolic syndrome), like a lack of physical activity. Indeed, the relationship between physical exercise and functional improvement has catched the attention of the scientific community, which is testing different approaches in healthy subjects and patients with psychotic disorders. The benefits of physical activity are described in patients with SCZ on weight, metabolic syndrome, and cardiovascular risk ; however, physical activity is too little invested in or quickly abandoned. Adapted physical activity (APA) is particularly indicated in psychiatry, and the benefits of APA in patients with SCZ is proven.

The enriched environment (EE) consists of a set of behavioral interventions to maximize stimulations, which can rely on Virtual Reality (VR) technologies. An immersive, realistic, and attractive environment will increase motivation and observance. Furthermore, the training is safer and more controlled than in outdoor conditions. A research combining EE and VR has used stationary bikes connected to a screen to maintain the physical, cognitive, and social capabilities of elderly subjects. To our knowledge, there are no studies using an EE with VR for the practice of APA in patients suffering from a FEP. However, this EE could lead, with its playful and immersive aspect, to a better observance to APA.

An adapted physical activity program usig connected bike with enriched environment (DYNAMO-PSYProgram) could help to prevent weight gain et metabolic syndrome in a population of First Episode Psychosis patients treated with antipsychotic drugs.

This study is a prospective, monocentric PILOT study. The main objective will be to check that at least 70% of the patients can complete the 20 sessions of the program.

Methods

The treatment being studied involves a program (DYNAMO-PSY) of adapted physical activity with an enriched environment (connected bike, visualized and experienced roads in virtual reality) and supervised, with (on average) two sessions per week, a total of 20 sessions to be completed over a maximum of 15 weeks. The usual hygienic-dietetic care is not modified by the study and consists of the care proposed to patients of the GHU Paris Psychiatry and Neuroscience who have had a first psychotic episode and are treated primarily with medication: clinical and biological monitoring

The visits planned by the experimental protocol include:

* a pre-inclusion visit V0, where oral and written information about the study is given to the patient by one of the study investigators
* an inclusion visit = V1 (at least 48 hours after V0, and no more than 15 days later, so that the patient has time to consider participating in the study), with the signing of the informed consent form in the presence of a study investigator.
* an end-of-study visit (= V2), 15 weeks after the inclusion visit V1.

The following elements will be collected for all patients at V1 :

* age, sex at birth, gender
* patients sports habits (weekly physical activity duration, type of physical activity), presence or absence of a dietary follow-up, current psychotropic medication, substance use will also be collected.

The following elements will be collected for all patients at V1 and V2 :

* psychiatric symptomes, with CAARMS, PANSS, HAD-A, HAD-D, SNS, STAI A / B.
* self-esteem measured by Rosenberg self-esteem scale (RSES)
* functional impact with the WHO-QOL-BREF (World Health Organization-Quality Of Life) quality of life questionnaire, the SOFAS, and the general functioning score on the Global Assessment of Functioning (GAF) scale
* cognitive tests : Memory with scores at California Verbal Learning Test (CVLT), digit span, Corsi Block, MEM-III, Executive functions with Trail Making Test (TMT), verbal fluencies, Stroop test, 'test des comissions', autoquestionnaire Behavior Rating Inventory of Executive Function (BRIEF) Processing speed with scores at Coding Test and Symbol search. Attention with score at Symbol Searchn coding D2R task.
* adherence to antipsychotic treatment with the MARS (Medication Adherence Rating Scale) questionnaire.

The following cardiometabolic parameters will be recorded at V1 and V2:

* weight (in kg, assessed with a bioimpedance scale)
* body mass index (weight / height^2)
* waist circumference (in cm, measured with a tape measure)
* fasting blood glucose concentration (in mmol/l)
* blood triglyceride levels (mmol/l)
* cholesterol levels (total, HDL, LDL)
* systolic and diastolic blood pressure (in mmHg)

Outcomes :

Primary Outcome is to calculate the proportion of patients who fully complete the DYNAMO-PSY program.

It will be measured by the Completion rate : ie. the number of patients who fully complete the DYNAMO-PSY program.

The completition rate to the DYNAMO-PSY program is calculated as the proportion: number of patients who completed the program / number of patients included in the study.

Secondary Outcomes :

1. Explore the acceptability and compliance to the DYNAMOPSY program, which will be evaluated with :

   * Acceptability rate (number of patients accepting the program / number of eligible patients)
   * compliance rate (number of sessions completed / number of planned sessions).
   * The mean duration of the program.
2. Explore effect of DYNAMOPSY program on psychiatric symptomes (scores at CAARMS, PANSS, HAD-A, HAD-D, and SNS), cognition (memory with scores at CVLT, number memory, corsi task, executive functions with TMT, fluencies, stroop test, 'test des comissions', BRIEF, attention with score at D2R), general status (self-esteem with WHO-QOL-BREF, quality of life with SOFAS, level of functioning scores with GAF), adhesion to antipsychotic treatment (MARS Scale) between V1 and V2.
3. Explore the effect of DYNAMOPSY program on cardiometabolic parameters (weight, body mass index, waist circumference, fasting blood glucose concentration, blood triglyceride levels, cholesterol levels, systolic and diastolic levels (HDL, LDL, total), systolic and diastolic blood presure.
4. Explore the influence of age, sex, sports habits, presence of a dietary follow up, current psychotropic medication, substance use on completing the program.

Statistics :

Statistical analysis will be performed

Sample size :

The sample size was estimated using the confidence interval approach for a proportion (Clopper-Pearson exact test). It is considered that the minimum compliance rate (patients who complete the program/adherent patients) for planning the main study should be at least 70%. Therefore, given the pilot nature of the study, the confidence level (1-alpha) is set at 80% and a bilateral confidence interval equal to 0.18 (CI=0.70-0.88), a necessary sample size of 40 subjects was estimated.

All continuous variables, including changes from baseline, will be summarized with the following statistics:

* Mean
* Standard deviation
* 95% confidence interval
* Median
* Interquartile range (IQR) for asymmetric variables Missing values will be indicated.

The following formulas will be used, depending on how the post-baseline endpoint is defined, for each planned visit and for each time point where both baseline and post-baseline values are available:

* Change from baseline = post-baseline value - baseline value
* Percentage change from baseline = (post-baseline value - baseline value) / baseline value * 100%
* Ratio to baseline = post-baseline value / baseline value

Baseline characteristics: An initial descriptive analysis will be performed for all collected variables, including :

* For all quantitative variables:

  * Absolute, relative, and cumulative frequency
  * 95% confidence interval
  * Interquartile range
  * Indication of missing values
* For all qualitative variables:

  * Absolute, relative, and cumulative frequency
  * 95% confidence interval
  * Indication of missing values

For the evaluation of the primary objective, the percentage of patients who completed the DYNAMO-PSY program according to the protocol will be calculated based on the specified criteria in the primary objective:

• The DYNAMO-PSY program is considered completed when the patient has completed all 20 sessions for a duration of up to 15 weeks.

The hypothesis assumes a non-inferior completion rate of 70%. A 95% confidence interval around the percentage of patients who completed the program will be provided.

Secondary objectives:

1. For acceptance rate (number of patients accepting the program / number of eligible patients) and compliance rate (number of completed sessions / number of planned sessions), the percentage and 95% confidence interval will be provided.
2. Regarding the comparison of psychiatric symptoms, general status (self-esteem, quality of life, overall functioning), neurocognition, cardiometamolic parameters before and after the DYNAMO-PSY program, the following exploratory analyses will be conducted:

   * Quantitative data will be compared between completers and non-completers using Student's t-tests or ANOVA, or non-parametric tests (Wilcoxon, Mann-Whitney, Kruskal-Wallis) if the distribution remains asymmetric even after appropriate transformation (e.g., Tukey's power transformation scale).
   * Paired tests will be used for comparing repeated measurements within the same patients.
   * Qualitative data will be compared using Chi-squared tests or Fisher's exact tests for independent groups, and McNemar's tests for paired groups (repeated measurements).
3. The influence of age, sex, current psychotropic medication, substance use, dietery follow up, sport habbit on completing the program will be analyzed with chi square tests.

ELIGIBILITY:
Inclusion Criteria:

- Patient suffering or having suffered from a FEP, corresponding to the criteria of brief psychotic episode or schizoaffective disorder in the DSM-5, within the last two years.

Or suffering from schizophrenia or a schizoaffective disorder, evolving for less than two years.

* Aged 18 to 30 years.
* Male or female.
* inpatient or outpatient.
* Treated with antipsychotic (typical or atypical).
* Willing to participate in the study and having signed the informed consent form after oral and written information.
* Affiliated or beneficiary of a health insurance scheme.

Exclusion Criteria:

* Patient not fluent in French.
* Patient in detention or under protective measures.
* Patient hospitalized without consent
* Medical contraindication to cycling (notably ventricular arrhythmia, or prolonged QT interval), validated by a medical opinion.
* Known epilepsy.
* Pregnant or breastfeeding women.

Specific Contraindications to Virtual Reality:

* High susceptibility to motion sickness.
* Vestibular disorders.
* Anomalies in postural statics and/or dynamic balance with proprioception disorders.
* Uncorrected ocular or oculomotor disorders.
* Frequent migraines.
* Severe anxiety

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Completion rate of the DYNAMO-PSY program | From enrollment to the end of the program at 15 weeks
  The main objective will be to assess the completion rate of the dynamopsy program.
  Then, the primary outcome measure will be the completion of the program by the participant (Yes/No).
  For each patient included in the study, the number of sessions completed will be recorded. The DYNAMO-PSY program consists of 20 sessions in total. The DYNAMO-PSY program is considered completed when the patient has completed 20 sessions (otherwise, the program is considered abandoned).
  The completion rate to the DYNAMO-PSY program will be calculated as the proportion : number of patients who completed the program / number of patients included in the study.

SECONDARY OUTCOMES:
Social and Occupational Functioning | at enrollment and at 15 weeks
  Total score at SOFAS (Social and Occupational Functioning Assessment Scale)
Global Functionning | at enrollment and at 15 weeks
  Total score at Global Assessment of Functioning (GAF) scale
Executive functions - Inhibition | at the enrollment and at 15 weeks
  Score at Stroop Test
Executive functions : Cognitive flexibility | at the enrollment and at 15 weeks
  Score at Trail Making Test
Executive functions - symptoms inventory | at the enrollment and at 15 weeks
  Composite executive globale Score (CEG) at the BRIEF questionnaire ( Behavior Rating Inventory of Executive Function ). Questionnaire fulfilled by the patient himself.
Memory : Digit Span | at enrollment and at 15 weeks
  Total score at Digit Span task
Memory : visuospatial working memory | at enrollment and at 15 weeks
  Total score at Corsi block - taping task
Memory : Episodic memory | at enrollment and at 15 weeks
  Total Score at MEM III task
Memory : Processing speed (visual perception) | at enrollment and at 15 weeks
  Total score at Symbol Search task
Attention | at enrollment and at 15 weeks
  Total score at D2R task
Adherence to antipsychotic treatment | at enrollment and at 15 weeks
  Total score at MARS (Medication Adherence Rating Scale) autoquestionnaire
Weight | at enrollment and at 15 weeks
  Weight (in kg, assessed with a bioimpedance scale)
Body mass index | at enrollment and at 15 weeks
  Calculated as : weight / height^2
waist circumference | at enrollment and at 15 weeks
  in cm, measured with a tape measure
fasting blood glucose concentration | at enrollment and at 15 weeks
  fasting blood glucose concentration (in mmol/l)
blood triglyceride levels | at enrollment and at 15 weeks
  blood triglyceride levels (mmol/l)
Total cholesterol level | at enrollment and at 15 weeks
  Total cholesterol blood level in mmol/L
HDL cholesterol level | at enrollment and at 15 weeks
  HDL cholesterol blood level in mmol/L
LDL cholesterol level | at enrollment and at 15 weeks
  LDL cholesterol blood level in mmol/L
Systolic blood pressure | at enrollment and at 15 weeks
  Systolic blood pressure in mmHg
diastolic blood pressure | at enrollment and at 15 weeks
  diastolic blood pressure in mmHg
Quality of life as assessed by WHO-QOL-BREF | at enrollment and at 15 weeks
  Total Score at WHO-QOL-BREF (World Health Organization-Quality Of Life) questionnaire
Psychotic symptomes as measured with the PANSS | at the enrollment and at 15 weeks
  Psychotic symptomes measured with the PANSS (Positive and negative symptomes scale).
  We will measure three outcomes :
  * Positive symptomes : total score at the positive symptomes subscale of the PANSS
  * Negative symptomes : total score at the positive symptomes subscale of the PANSS
  * General symptomes : total score at the general symptomes subscale of the PANSS
Memory - Verbal Learning | at enrollment and at 15 weeks
  Total score at California Verbal Learning Test (CVLT)
Executive functions Verbal fluencies | at the enrollment and at 15 weeks
  Total score at verbal fluencies task
Acceptibility rate of the DYNAMO-PSY program | From enrollment to the end of the program at 20 weeks
  We will calculate the acceptibility rate as followed :
  Number of patients included / number of eligible patients
Compliance of participants to the DYNAMO-PSY program | From enrollment to the end of the program at 15 weeks
  For each participants, we will measure how many sessions have been completed.
  The compliance rate will be measured as followed :
  Number of sessions completed by the participant / 20 (number of planned sessions)
Negative psychotic symptoms as measured by SNS | at enrollment and at 15 weeks
  Total score at self evaluation of negative symptoms scale (autoquestionnaire).
Memory : Number memory | at the enrollment and at 15 weeks
  Score at number memory task
Executive functions : Planification | at the enrollment and at 15 weeks
  Score at the french test -test des comissions-
Depression symptomes as measured with HAD-D | at enrollment and at 15 weeks
  Score at the -depression- subscale of the HAD scale (autoquestionnaire)
Mean duration of the program | at the first and at the last session of the DYNAMO-PSY program
  For each participants that completed the DYNAMO-PSY program, we will measure time (in days) between the first and the last session (ie the 20th) of the DYNAMOPSY program.
  We will calculate the mean duration of the program among participants that completed the program.
Anxiety symptoms as measured by HAD-A | at enrollment and at 15 weeks
  Score at anxiety subscale of Hospital anxiety and depression scale (HAD-A) (autoquestionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Raphaëlle LEROUX AUGER, DR, Principal Investigator — Pôle PEPIT - Centre d évaluation pour Jeunes Adultes et Adolescents (CJAAD)